CLINICAL TRIAL: NCT02789436
Title: Effect of Probiotic Lactobacillus Reuteri-containing Lozenges (Prodentis) on Halitosis in Patients With Chronic Periodontitis
Brief Title: Effect of Probiotic Lozenges on Halitosis in Patients With Chronic Periodontitis
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Zagreb (Other)
Collaborators: BioGaia AB (Industry)
Responsible Party: Principal Investigator, Larisa Musić, Doctor of Dental Medicine, University of Zagreb
Allocation: Randomized | Model: Parallel | Masking: Double
Other Study IDs: 05-PA-26-10/15
Record Dates: First submitted 2016-04-04; First posted 2016-06-03 (Estimated); Last update posted 2016-06-03 (Estimated); Status verified 2016-05

CONDITIONS: Halitosis
Keywords: halitosis; chronic periodontitis; probiotic
MeSH Terms: conditions — Halitosis; Chronic Periodontitis

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- L. reuteri Prodentis® lozenges (Experimental): 15 subjects
  Probiotic lozenges used in the trial is a non-commercial product provided by BioGaia AB, Lund, Sweden. The Probiotic lozenges consist of a minimum of 200 million live L. reuteri (L. reuteri DSM 17938 and L. reuteri ATCC PTA 5289 (L. reuteri Prodentis®). Probiotic lozenges are used twice daily for 28 days.
  Interventions: Drug: L. reuteri Prodentis® lozenges
- Placebo lozenges (Placebo Comparator): 15 subjects
  Placebo lozenges used in the trial is non-commercial product provided by BioGaia AB, Lund, Sweden.Placebo lozenges are taken twice daily for 28 days.
  Interventions: Other: Placebo lozenges

INTERVENTIONS:
Drug: L. reuteri Prodentis® lozenges — Twice daily, for 28 days
  Arms: L. reuteri Prodentis® lozenges
Other: Placebo lozenges — Twice daily, for 28 days
  Arms: Placebo lozenges

SUMMARY:
The purpose of this study is to determine whether Lactobacillus reuteri-containing lozenges (Prodentis) are effective in treatment of halitosis in patients with chronic periodontitis.

DETAILED DESCRIPTION:
Bad breath (oral malodor, lat. halitosis) is amongst most common patients' complaints in the dental office. Ironically, available literature and research done on this topic thus far are relatively scarce. Oral malodor is most commonly caused by oral bacteria (87%), yet it can also be sourced from ear, nose and throat region and in a small percentage from distant parts of the body or is of unknown origin. Periodontal pathogens and other Gram(-) anaerobic microorganisms such as Porphyromonas gingivalis, Treponema denticola, Prevotella intermedia, Fusobacterium nucleatum, Enterobacter cloacae, Prevotella loescheii and Porphyromonas endodontalis are regarded as producers of malodorous gases. Namely, these bacterial species and periodontal pathogens particularly produce so called volatile sulfur compounds (VSC) which give mouth air its malodorness. Methylmercaptan, hydrogen sulfide and dimethyl sulfide are waste products of bacterial metabolism, specifically degradation of sulfur-, methionine- and cysteine-containing aminoacids. Offensive smells also stem from other compounds which do not contain sulfur, diamines and polyamines such as cadaverine, putrescine and skatole.

Probiotics are defined as living microorganisms which are considered to have beneficial health effect on their host when consumed in adequate amount. Regarding their advantageous role in periodontal disease, inhibition of specific periodontal pathogens and alteration of host immune response through multifactorial causes are thought to be their main working mechanisms. Reuterin and reutericyclin are two bacteriocins produced by Lactobacillus reuteri that inhibit growth of pathogenic bacteria, while bacterium also exhibits strong capacity of host tissue adherence and subsequent competition with pathogens.

Based on this data, research on efficacy of probiotic lozenges on halitosis in patients with chronic periodontitis.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients, above age of 30
* Non-smokers or ex-smokers (not smoking in the past year)
* Moderate to advanced untreated chronic periodontitis
* Good compliance and following of oral hygiene instructions
* Halitosis in active phase and patient's subjective complaint
* Informed consent by the patient

Exclusion Criteria

* Aggressive periodontitis
* Antibiotics administered up to 3 months prior to this study
* Pregnancy and breastfeeding
* Immunosuppressive therapy
* Oral neoplasms (including radiation or chemotherapy)
* Diabetes mellitus
* Acute oral inflammation or infection
* Poor, unsatisfactory oral hygiene and lack of compliance
* Use of dietary supplements containing probiotics within 2 weeks prior to study start

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2016-06; Primary Completion 2016-09 (Estimated)

PRIMARY OUTCOMES:
Change in VSC concentration in mouth air | 28 days
  Assessed with halimeter

SECONDARY OUTCOMES:
Changes in halitosis associated quality of life | 28 days
  Assessed with Halitosis Associated Life-quality Test (Kizhnev et al., 2011)
Change from Baseline in Plaque Accumulation (PCR) | 28 days
  Assessed with PCR index (Plaque Control Record - O'Leary et al., 1972)
Change from Baseline in Bleeding on Probing (BOP) | 28 days
  Assessed with BOP index (Bleeding on Probing, Ainamo and Bay, 1975)

CONTACTS AND LOCATIONS:
Overall Officials: Darije Plančak, Professor, Study Director — University of Zagreb
Locations (1):
- University of Zagreb, School of Dental Medicine Zagreb, Zagreb, Croatia

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Loesche WJ, Kazor C. Microbiology and treatment of halitosis. Periodontol 2000. 2002;28:256-79. doi: 10.1034/j.1600-0757.2002.280111.x. PMID 12013345
- [Background] Delanghe G, Ghyselen J, van Steenberghe D, Feenstra L. Multidisciplinary breath-odour clinic. Lancet. 1997 Jul 19;350(9072):187. doi: 10.1016/S0140-6736(05)62354-9. No abstract available. PMID 9250193
- [Background] Persson S, Claesson R, Carlsson J. The capacity of subgingival microbiotas to produce volatile sulfur compounds in human serum. Oral Microbiol Immunol. 1989 Sep;4(3):169-72. doi: 10.1111/j.1399-302x.1989.tb00246.x. PMID 2639302
- [Background] Persson S, Edlund MB, Claesson R, Carlsson J. The formation of hydrogen sulfide and methyl mercaptan by oral bacteria. Oral Microbiol Immunol. 1990 Aug;5(4):195-201. doi: 10.1111/j.1399-302x.1990.tb00645.x. PMID 2082242
- [Background] Goldberg S, Kozlovsky A, Gordon D, Gelernter I, Sintov A, Rosenberg M. Cadaverine as a putative component of oral malodor. J Dent Res. 1994 Jun;73(6):1168-72. doi: 10.1177/00220345940730060701. PMID 8046106
- [Background] Walker WA. Mechanisms of action of probiotics. Clin Infect Dis. 2008 Feb 1;46 Suppl 2:S87-91; discussion S144-51. doi: 10.1086/523335. PMID 18181730
- [Background] Haukioja A. Probiotics and oral health. Eur J Dent. 2010 Jul;4(3):348-55. PMID 20613927